CLINICAL TRIAL: NCT04365166
Title: Study of Clinical and Immune Severity Profiles of Patients Infected With SARS-Cov2
Brief Title: Study of Clinical and Immune Severity Profiles of Patients Infected With SARS-Cov2 (COVID-19)
Acronym: REACOVIM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-COVID19-05; 2020-A00898-31 (Other: IDRCB)
Record Dates: First submitted 2020-04-19; First posted 2020-04-28 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Respiratory Tract Infections; Respiratory Tract Disease
MeSH Terms: conditions — Respiratory Tract Infections; Respiratory Tract Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological samples include:
  * blood
  * urine
  * nasopharyngeal swab
  * tracheal suction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The SARS-CoV2 virus causes severe or even fatal disease in a fraction of infected people. The clinical severity is based on a complicated pneumopathy with acute respiratory distress syndrome that can lead to multi-visceral failure. The underlying mechanism is a cytokinergic storm, an emerging facet of immunological dysregulation.

This clinical trial is aimed to understand the mechanisms of this immunological dysregulation in order to identify therapeutic levers.

The main objective is to understand the relationships between clinical severity, death or morbidity of resuscitation management, and immune status (i.e., immune pathways activated or not). Immune status will be investigated at many levels of organization (i.e., circulating leukocytes, cytokines and chemokines, transcripts).

The secondary objectives are :

* to understand what is responsible for clinical severity, viral load, or immune activation;
* to highlight the consequences of immunological dysregulation on associated risks (i.e., immunosuppression leading to the emergence of infectious comorbidities) as well as the functioning of neurotransmission through metabolic pathway diversions. The impact of dysimmunity on these biological pathways will be assessed with a metabolomic analysis;
* to understand the mechanisms of vulnerability related to the field. Moreover, while co-morbidities are likely to be a risk factor for severe disease progression, there are many situations in which they do not occur. Stress, with its neurovegetative and endocrinological dimensions, modulates the immune response. It is essential to know whether the stress response plays a role in immunological dysregulation. This analysis is a prerequisite for understanding the conditions of treatment with glucocorticoids.

Angiotensin converting enzyme type 2 (ACE2) also plays a likely role in host viral infection. It is also thought to play an important role in the emergence of severe syndromes by affecting the quality of vascular response.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to intensive care unit with confirmed SARS-CoV2 infection
* Patient older than 18 years old

Exclusion Criteria:

* Patient coming from another intensive care unit after more than 5 days in the intensive care unit
* Known immunosuppression:

  * Known or suspected HIV
  * Known or suspected immunosuppression :
  * Organ transplantation
  * Marrow transplant
  * Congenital deficit
  * Received immunosuppressive therapy within 30 days (azathioprine, methotrexate, tacrolimus, cyclosporine, sirolimus, cyclophosphamide, rituximab, anti-TNF, JAK inhibitors, corticosteroids >10mg/day over the last 30 days, recent covid-19 corticosteroid therapy >1mg/kg prednisolone or equivalent >5 days)
  * Administration of chemotherapy within the last 3 months
* Current pregnancy or breastfeeding
* Patient under 18 years of age
* Incapacitated adults and persons deprived of their liberty
* Refusal by the patient or his/her support person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population is a population infected with SARS-CoV2 and justifying hospitalisation in an intensive care unit, i.e. presenting at least one immediate vital failure that would lead in short term to the death of the patient without the implementation of an adapted active therapeutic intervention. As the variable of interest is immuno-inflammatory activation, patients with an immune deficiency of any origin will be excluded. Patients will be recruited from patients admitted to the intensive care unit with biological confirmation of SARS-Cov2 infection.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-21 (Actual); Primary Completion 2022-04-21 (Estimated); Study Completion 2022-04-21 (Estimated)

PRIMARY OUTCOMES:
Mortality | 90 days following the enrollment
  Mortality
Immune response - Plasma cytokine profile | Through study completion (90 days following the enrollment)
  Th1/Th2/Th17/Treg balance, Type I Interferons and inflammation
Immune response - Phenotype of circulating cells | Through study completion (90 days following the enrollment)
  T cells (CD3, CD4, CD8, PD1, FAS, CD45RO, CTLA4+, CXCR5, CXCR3, CCR6, CD69, CD95, HLA-DR) and B cells (CD3, CD19, CD27, IgD, CD69) with cell subtypes and memory/naive compartments (CD27, CD38, IgD, IgG1, IgG2, IgG3, CD20, CD24), NK cells (CD14, CD16, CD56, HLA-DR), monocytes (CD14, CD45, HLA-DR, PDL-1)

SECONDARY OUTCOMES:
Severity criteria - Duration of stay in intensive care unit | 90 days following the enrollment
  Number of days in intensive care unit
Severity criteria - Duration of hospitalization stay | 90 days following the enrollment
  Number of days of hospitalization
Severity criteria - Duration of period out of hospital | 90 days following the enrollment
  Number of days out of hospital
Severity criteria - Duration without mechanical ventilation | 90 days following the enrollment
  Number of days without mechanical ventilation (invasive/non-invasive)
Severity criteria - Duration without ventilation | 90 days following the enrollment
  Number of days not being ventilated
Severity criteria - Duration without intubation | 90 days following the enrollment
  Number of days not being intubated
Severity criteria - Number of transfusions | 90 days following the enrollment
  Number of transfusions
Severity criteria - Duration of the period without cathecholamines | 90 days following the enrollment
  Number of days without cathecholamines
Severity criteria - Duration of the period without dialysis | 90 days following the enrollment
  Number of days without dialysis
Severity criteria - SOFA | Through study completion (90 days following the enrollment)
  Sepsis-related Organ Failure Assessment (SOFA) Score
Severity criteria - LIS | Through study completion (90 days following the enrollment)
  Lung Injury Score (LIS)
SARS-Cov2 viral load | Through study completion (90 days following the enrollment)
  SARS-Cov2 viral load will be measured in blood and in broncho-tracheal secretions
Emergence of concomitant infections | 90 days following the enrollment
  Co-infections and acquired infections (bacterial or fungal) in intensive care unit, in particular based on an all-site positive PCR for EBV and/or CMV and/or HSV
Emergence of concomitant infections - Phenotype of circulating cells | Through study completion (90 days following the enrollment)
  T cells (CD3, CD4, CD8, PD1, FAS, CD45RO, CTLA4+, CXCR5, CXCR3, CCR6, CD69, CD95, HLA-DR) and B cells (CD3, CD19, CD27, IgD, CD69) with cell subtypes and memory/naive compartments (CD27, CD38, IgD, IgG1, IgG2, IgG3, CD20, CD24), NK cells (CD14, CD16, CD56, HLA-DR), monocytes (CD14, CD45, HLA-DR, PDL-1)
Stress physiological profile - Sympathetic tone | Through study completion (90 days following the enrollment)
  Heart rate variability
Stress physiological profile - Temperature | Through study completion (90 days following the enrollment)
  Core temperature
Stress physiological profile - Glucocorticoids | Through study completion (90 days following the enrollment)
  Quantity of glucocorticoids in the urine during 24 hours and at night
Angiotensin converting enzyme type II (ACE2) polymorphism - ACE | At enrollment
  ACE Polymorphism
Angiotensin converting enzyme type II (ACE2) polymorphism - ACE2/ACE1 | At enrollment
  Protein expression of ACE2 vs. ACE1 and angiotensin II chain proteins
Comorbidities - diabetes | At enrollment
  Diabete diagnosis
Comorbidities - Heart disease | At enrollment
  Heart disease diagnosis
Comorbidities - organ failure | At enrollment
  Organ failure diagnosis
Plasma concentrations of several metabolic pathways - GABA | Through study completion (90 days following the enrollment)
  GABA level in blood and urine
Plasma concentrations of several metabolic pathways - Glucocorticoid | Through study completion (90 days following the enrollment)
  Glucocorticoid level in blood and urine
Plasma concentrations of several metabolic pathways - Tryptophan | Through study completion (90 days following the enrollment)
  Tryptophan in blood and urine
Plasma concentrations of several metabolic pathways - Serotonin | Through study completion (90 days following the enrollment)
  Serotonin level in blood and urine
Plasma concentrations of several metabolic pathways - Dopamin | Through study completion (90 days following the enrollment)
  Dopamin level in blood and urine
Plasma concentrations of several metabolic pathways - Cathecholamines | Through study completion (90 days following the enrollment)
  Catecholamines level in blood and urine
Plasma concentrations of several metabolic pathways - Arachidonic acid derivatives | Through study completion (90 days following the enrollment)
  Arachidonic acid derivatives level in blood and urine
Plasma concentrations of several metabolic pathways - Endocannabinoids | Through study completion (90 days following the enrollment)
  Endocannabinoids level in blood and urine

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Percy Military Teaching Hospital, Clamart
  - Bégin Military Teaching Hospital, Saint-Mandé